CLINICAL TRIAL: NCT01884441
Title: Phase II Study With Bendamustine, Gemcitabine and Vinorelbine (BeGEV) as Induction Therapy in Relapsed/Refractory Hodgkin's Lymphoma Patients Before High Dose Chemotherapy With Autologous Hematopoietic Stem Cells Transplant
Brief Title: Bendamustine, Gemcitabine and Vinorelbine (BeGEV) as Induction Therapy in Relapsed/Refractory Hodgkin's Lymphoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2010-002; 2010-022169-91 (EudraCT Number)
Record Dates: First submitted 2013-05-27; First posted 2013-06-24 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin; Lymphoma; refractory; relapsed
MeSH Terms: conditions — Hodgkin Disease; Lymphoma; Recurrence | interventions — Bendamustine Hydrochloride; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BeGEV (Experimental): Bendamustine, Gemcitabine and Vinorelbine (BeGEV)
  Interventions: Drug: Bendamustine; Drug: Gemcitabine; Drug: Vinorelbine

INTERVENTIONS:
Drug: Bendamustine — Schedule:
  Day 2: Bendamustine 90mg/mq Day 3: Bendamustine 90mg/mq for a maximum of 4 cycles
  Other Names: Ribomustin
Drug: Gemcitabine — Day 1: Gemcitabine 800mg/mq, Day 4: Gemcitabine 800mg/mq for a maximum of 4 cycles
  Other Names: Gemzar
Drug: Vinorelbine — Day 1 Vinorelbine 20mg/mq for a maximum of 4 cycles
  Other Names: Navelbine

SUMMARY:
Test of bendamustine in combination with gemcitabine and vinorelbine could contribute to a higher response rate with the reduction of toxic side effects

DETAILED DESCRIPTION:
The aim of this study is to evaluate bendamustine, gemcitabine and vinorelbine (BeGEV) scheme efficacy as induction therapy to high dose chemotherapy with Allogeneic Hematopoietic Stem-Cell Transplantation (AHSCT) for patients with relapsed/refractory Hodglin's Lymphoma (HL).

Four BeGEV courses repeated every 3 weeks in the absence of any reasons listed in the paragraph 7.5; whenever an objective response is observed at disease evaluation performed after IV cycle patients undergo to high dose chemotherapy with AHSCT (conditioning regimens based on preference of each Centre).

ELIGIBILITY:
Inclusion Criteria:

* relapsed/refractory disease after receiving one line of standard chemotherapy
* history of classical Hodgkin's Lymphoma (HL)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* at least one site of measurable nodal disease at baseline ≥ 1.5 cm
* Absolute Neutrophils Count (ANC) ≥ 1.5 x 109/L; Platelets count ≥ 75 x 109/L

Exclusion Criteria:

* Diagnosis of Nodular lymphocyte predominant Hodgkin's lymphoma (NLPHL)
* prior radiation therapy ≤ 3 weeks prior to start of study treatment
* any concurrent anti-cancer therapy
* evidence of another malignancy not in remission or history of such a malignancy within the last 2 years.
* aspartate aminotransferase (AST/SGOT) and/or alanine aminotransferase (ALT/SGPT) ≥ 2.5 x upper limit of normal (ULN) or ≥ 5.0 x ULN if the transaminase elevation is due to disease involvement
* known history of Human immunodeficiency virus (HIV)seropositivity
* hepatitis B virus (HBV) or hepatitis B virus (HCV)active hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 3 months
  response rate after BeGEV in terms of Complete Response (CR)evaluated by fludeoxyglucose Positron emission tomography (FDG-PET) and Computed Tomography (CT-scan) after four cycles.

SECONDARY OUTCOMES:
overall response rate | 3 months
  To assess the response rate after BeGEV in terms of overall response rate (ORR) =Complete Response (CR) plus Partial Response (PR)).
mobilization potential of the combination | 3 months
  To evaluate the mobilization potential of BeGEV.
toxicity of the combination | 3 months
  To evaluate the toxicity of BeGEV in terms of haematological and extra-haematological side effects according to CTCAE definitions v 3.0.
Progression free survival (PFS), Overall Survival (OS). | 2 years
  Progression free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

REFERENCES:
- [Derived] Santoro A, Mazza R, Pulsoni A, Re A, Bonfichi M, Zilioli VR, Zanni M, Merli F, Anastasia A, Luminari S, Annechini G, Gotti M, Peli A, Liberati AM, Di Renzo N, Castagna L, Giordano L, Ricci F, Carlo-Stella C. Five-year results of the BEGEV salvage regimen in relapsed/refractory classical Hodgkin lymphoma. Blood Adv. 2020 Jan 14;4(1):136-140. doi: 10.1182/bloodadvances.2019000984. PMID 31935284
- [Derived] Santoro A, Mazza R, Pulsoni A, Re A, Bonfichi M, Zilioli VR, Salvi F, Merli F, Anastasia A, Luminari S, Annechini G, Gotti M, Peli A, Liberati AM, Di Renzo N, Castagna L, Giordano L, Carlo-Stella C. Bendamustine in Combination With Gemcitabine and Vinorelbine Is an Effective Regimen As Induction Chemotherapy Before Autologous Stem-Cell Transplantation for Relapsed or Refractory Hodgkin Lymphoma: Final Results of a Multicenter Phase II Study. J Clin Oncol. 2016 Sep 20;34(27):3293-9. doi: 10.1200/JCO.2016.66.4466. Epub 2016 Jul 5. PMID 27382096